CLINICAL TRIAL: NCT03498794
Title: Internal Ureteral Stent Versus Percutaneous Nephrostomy Tube in Management of Acutely Obstructed Infected Kidney in the Presence Upper Urinary Tract Stones: A Prospective, Randomized Study
Brief Title: Ureteral Stent Versus Percutaneous Nephrostomy in Acutely Obstructed Infected Kidney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MMMohammed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: US VS PCN
Record Dates: First submitted 2018-03-02; First posted 2018-04-17 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Management of Obstructed Infected Kidney

STUDY DESIGN:
Intervention Model Description: Comparison Between Ureteral Stent versus Percutaneous Nephrostomy in Obstructed infected kidney due to Ureteric calculi
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ureteral stent (Active Comparator): Technique of ureteral stent insertion:
  All patients will be in lithotomy position, and an endoscopy operating table with fluoroscopic imaging capability will be used. Before the procedures, all patients will have retrograde ureteropyelography. Then, a 0.035-inch hydrophilic guide wire will be placed into the renal pelvis under the guidance of flexible cystoscope.
  The ureteral stent will be inserted retrograde by using flexible cystoscope, under mild sedation or local anesthesia by instilling 2% xylocain gel per urethra. Patients will be covered by specific antimicrobial therapy according to urine and/or blood culture. This treatment will be continued until there was no fever and any evidence of infection disappeared. A Foley's catheter will be left in the bladder for 2 hours in all patients. In each case the type of stent will be that of 5 or 6 F, with side-holes and remain in place until definitive treatment of stone.
  Interventions: Procedure: Ureteral stent
- Percutaneous nephrostomy tube (Active Comparator): Technique of PCN insertion:
  Percutaneous nephrostomy will be performed in the angiography suite by a urologist with the patient under local anesthesia. All the patients will be given non-nephrotoxic antibiotics pre-operatively. The patients will be placed on the ultrasound table with fluoroscopic imaging capability in prone position and a pillow placed under the abdomen on the affected side to support the kidney. Then the initial puncture site will be chosen, cleaned and draped. Local anesthesia was injected and a stab incision was given at the puncture site. The 18-gauge Chiba needle will be inserted at the renal angle or at the posterior axillary line under ultrasound guidance into dilated pelvicalyceal system. Urine or pus drained out spontaneously or will be sucked with a disposable syringe and sample was sent to the laboratory for culture and sensitively.
  Interventions: Procedure: Ureteral stent

INTERVENTIONS:
Procedure: Ureteral stent — Patients will be randomized into 2 groups:
  Group (A): 75 patients with the use of ureteral stent. Group (B): 75 patients with the use of PCN.
  How the technique will be applied?
  Technique of ureteral stent insertion:
  The ureteral stent will be inserted retrograde by using flexible cystoscope.
  Technique of PCN insertion:
  Percutaneous nephrostomy will be performed in the angiography suite by a urologist with the patient under local anesthesia. All the patients will be given non-nephrotoxic antibiotics pre-operatively.
  Other Names: Percutanous nephrostomy tube

SUMMARY:
Non-malignant causes of ureter obstruction can be intrinsic such as stone disease, ureter stricture or congenital ureteropelvic junction obstruction, or extrinsic such as idiopathic retro peritoneal fibrosis. Nearly all clinicians agree that obstructing stones, with a concern for sepsis require immediate decompression of the urinary system.

Though large epidemiologic studies of the management of obstructed infected nephrolithiasis demonstrate higher rates of sepsis and mortality associated with PCN placement relative to ureteral stenting, the observational nature of the analysis highlights the need for prospective analyses of PCN vs stenting for obstructive nephrolithiasis.

Despite this obvious need, there are few studies comparing the efficacy of ureteral stenting vs PCN in the setting of obstructive urolithiasis. The choice between PCN and stenting is often made by the urologist at initial presentation and can be influenced by factors including disease severity, stone size, location of stone, eventual modality of definitive stone management, or even availability of in-house interventional radiology services.

Retrospective studies reveal that both procedures have high success rates. In the setting of unsuccessful stenting, PCN is often successful, but the contrary is not always true. Furthermore, patients are often selected for PCN over ureteral stenting in the setting of larger stones and if they are more severely ill.

Goldsmith et al studied 130 patients who underwent decompression for obstructing ureteral stone with PCN or stent placement. Although patients who underwent PCN placement had longer hospital stay, other outcomes such as time to definitive stone management, rates of spontaneous stone passage, and initiation of stone metabolic workup were not statistically different. The authors noted that the method of initial decompression correlated with eventual approach selected for definitive stone management. Patients treated with PCN were more likely to undergo percutaneous definitive management, while patients managed with ureteral stenting were more likely to be treatked with a ureteroscopic approach.

Two prospective studies comparing PCN vs stent management of obstructing ureteral stones have conflicting outcomes. Mokhmalji et al 6 in 2001 prospectively randomized 40 patients to receive either PCN or stent. Sixteen out of twenty stents were successfully placed while all twenty PCNs were successfully placed initially. All unsuccessful stents were successfully managed by PCN. Their results demonstrated that stent utilization was less successful as compared to PCN and there was a trend for longer antibiotic therapy due to persistent signs of urinary tract infection in patients who underwent stent placement.

In contrast, Pearle et al randomized 42 patients to receive PCN vs stents. This study failed to demonstrate one procedure to be more successful than the other. All 21stents and 20 out of 21 PCNs were successfully placed. One failed PCN successfully underwent stent placement. Their results demonstrated an increased incidence of bacterial urinary colonization post-procedure in the PCN group as compared to the stent group, but overall no differences in time to clinical improvement or length of stay were noted.

DETAILED DESCRIPTION:
Preoperative preparation:

* History taking: complete history will be taken, including personal, past and medical history as UTI.
* Examination: Included General examination (BMI will be estimated), abdominal, and neurological examination.
* Laboratory investigations:

  * Complete urine analysis: Physical, chemical and microscopic.
  * Urine culture at time of insertion.
  * Complete blood count (CBC).
  * Renal function test.
* Radiological evaluation:

  * Abdominal ultrasonography.
  * Plain KUB.
  * Non-contrast CT (NCCT-KUB).

How the technique will be applied?

Technique of ureteral stent insertion:

All patients will be in lithotomy position, and an endoscopy operating table with fluoroscopic imaging capability will be used. Before the procedures, all patients will have retrograde ureteropyelography. Then, a 0.035-inch hydrophilic guide wire will be placed into the renal pelvis under the guidance of flexible cystoscope.

The ureteral stent will be inserted retrograde by using flexible cystoscope, under mild sedation or local anesthesia by instilling 2% xylocain gel per urethra. Patients will be covered by specific antimicrobial therapy according to urine and/or blood culture. This treatment will be continued until there was no fever and any evidence of infection disappeared. A Foley's catheter will be left in the bladder for 2 hours in all patients. In each case the type of stent will be that of 5 or 6 F, with side-holes and remain in place until definitive treatment of stone.

Technique of PCN insertion:

Percutaneous nephrostomy will be performed in the angiography suite by a urologist with the patient under local anesthesia. All the patients will be given non-nephrotoxic antibiotics pre-operatively. The patients will be placed on the ultrasound table with fluoroscopic imaging capability in prone position and a pillow placed under the abdomen on the affected side to support the kidney. Then the initial puncture site will be chosen, cleaned and draped. Local anesthesia was injected and a stab incision was given at the puncture site. The 18-gauge Chiba needle will be inserted at the renal angle or at the posterior axillary line under ultrasound guidance into dilated pelvicalyceal system. Urine or pus drained out spontaneously or will be sucked with a disposable syringe and sample was sent to the laboratory for culture and sensitively. Then soft end of floppy J guide wire will be passed through the needle and needle was removed. The tract was dilated with Teflon facial dilators more than the diameter of the nephrostomy tube. After tract dilation a pig tail nephrostomy tube or a feeding tube of 8 Fr will be passed over the guide wire into the collecting system and secured with silk no.1. All patients were maintained on antibiotic prophylaxis after culture sample.

Operative evaluation:

* Operative time in minutes.
* Fluoroscopy time in seconds.
* Urine culture.
* Use of analgesics.
* Success of insertion.

Post operative evaluation (every week until definitive treatment of stone):

* Time to normal temperature 37.4C or less.
* Time to normal white blood count WBC of 10,000/mm.3 or less.
* Time to normal serum chemistry in case of uremic cases.
* Urine culture.
* length of hospital stay in days.
* Duration of diversion, The time until definitive stone treatment and specific treatment modality
* Duration of intravenous administration of antibiotics for high temperature)
* Quality of life (questionnaire immediately and 2 to 4 weeks postoperatively).
* The time until definitive stone treatment and specific treatment modality
* Complications were noted in immediate post-operative period and on follow up: Procedural failure, Injury to adjacent organs, Fever & Septicemia, Bleeding/Hematuria Painful Trigone irritation, PCN dislodgement or blockage, Ureteral Perforat;ion , Stent Migration, Stent Encrustation or Stone formation

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients with infected hydronephrosis.
2. Infected hydronephrosis due to ureteric stone or ureteric stricture.
3. Uremic and non uremic patients.

Exclusion Criteria:

* Patients with a contraindication to either form of drainage (uncorrected coagulopathy, urethral stricture disease, bladder outlet obstruction, pregnancy, ureteral stone greater than 15 mm., or Steinstrasse).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Ureteral stent vs percutaneous nephrostomy (PCN) for drainage obstructed infected kidney | 2 years from April 2018 to may 2020
  To compare between Ureteral stent versus Percutaneous Nephrostomy tube (PCN) in management of obstructed infected kidney by Improvement of infection clinically by decreasing high body temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud magdy, Asyut, Egypt

REFERENCES:
- [Background] Lynch MF, Anson KM, Patel U. Current opinion amongst radiologists and urologists in the UK on percutaneous nephrostomy and ureteric stent insertion for acute renal unobstruction: Results of a postal survey. BJU Int. 2006 Dec;98(6):1143-4. doi: 10.1111/j.1464-410X.2006.06513.x. No abstract available. PMID 17125470
- [Background] Sammon JD, Ghani KR, Karakiewicz PI, Bhojani N, Ravi P, Sun M, Sukumar S, Trinh VQ, Kowalczyk KJ, Kim SP, Peabody JO, Menon M, Trinh QD. Temporal trends, practice patterns, and treatment outcomes for infected upper urinary tract stones in the United States. Eur Urol. 2013 Jul;64(1):85-92. doi: 10.1016/j.eururo.2012.09.035. Epub 2012 Sep 25. PMID 23031677
- [Background] Ahmad I, Saeed Pansota M, Tariq M, Shahzad Saleem M, Ali Tabassum S, Hussain A. Comparison between Double J (DJ) Ureteral Stenting and Percutaneous Nephrostomy (PCN) in Obstructive Uropathy. Pak J Med Sci. 2013 May;29(3):725-9. doi: 10.12669/pjms.293.3563. PMID 24353616
- [Background] Goldsmith ZG, Oredein-McCoy O, Gerber L, Banez LL, Sopko DR, Miller MJ, Preminger GM, Lipkin ME. Emergent ureteric stent vs percutaneous nephrostomy for obstructive urolithiasis with sepsis: patterns of use and outcomes from a 15-year experience. BJU Int. 2013 Jul;112(2):E122-8. doi: 10.1111/bju.12161. PMID 23795789
- [Background] Yoshimura K, Utsunomiya N, Ichioka K, Ueda N, Matsui Y, Terai A. Emergency drainage for urosepsis associated with upper urinary tract calculi. J Urol. 2005 Feb;173(2):458-62. doi: 10.1097/01.ju.0000150512.40102.bb. PMID 15643207
- [Background] Mokhmalji H, Braun PM, Martinez Portillo FJ, Siegsmund M, Alken P, Kohrmann KU. Percutaneous nephrostomy versus ureteral stents for diversion of hydronephrosis caused by stones: a prospective, randomized clinical trial. J Urol. 2001 Apr;165(4):1088-92. PMID 11257644
- [Background] Pearle MS, Pierce HL, Miller GL, Summa JA, Mutz JM, Petty BA, Roehrborn CG, Kryger JV, Nakada SY. Optimal method of urgent decompression of the collecting system for obstruction and infection due to ureteral calculi. J Urol. 1998 Oct;160(4):1260-4. PMID 9751331